CLINICAL TRIAL: NCT03427996
Title: Evaluation of Effectiveness and Safety of Rotational Atherectomy in Routine Clinical Practice; A Multicenter, Prospective Observational Study
Brief Title: Evaluation of Effectiveness and Safety of Rotational Atherectomy in Routine Clinical Practice
Acronym: IRIS-ROTA
Status: Recruiting | Type: Observational
Sponsor: Seung-Jung Park (Other)
Collaborators: CardioVascular Research Foundation, Korea (Other)
Responsible Party: Sponsor-Investigator, Seung-Jung Park, Professor, Division of Cardiology, Asan Medical Center
Organization: Asan Medical Center (Other)
Other Study IDs: AMCCV2018-02
Record Dates: First submitted 2018-02-05; First posted 2018-02-09 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Atherosclerosis, Coronary; Coronary Stenosis
Keywords: rotational atherectomy
MeSH Terms: conditions — Coronary Artery Disease; Coronary Stenosis | interventions — Atherectomy, Coronary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Coronary disease
  Interventions: Procedure: Rotational atherectomy

INTERVENTIONS:
Procedure: Rotational atherectomy — Percutaneous coronary intervention with rotational atherectomy

SUMMARY:
This study evaluates the effectiveness and safety rotational atherectomy in routine clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 19 years old
* Patients who received rotational atherectomy
* The patient or guardian agrees to the study protocol and the schedule of clinical follow-up and provides informed, written consent, as approved by the appropriate Institutional Review Board/Ethics Committee of the respective clinical site.

Exclusion Criteria:

* Life expectancy <1y

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive percutaneous coronary intervention patients receiving rotational atherectomy
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2018-09-04 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2034-12-31 (Estimated)

PRIMARY OUTCOMES:
Target vessel failure (TVF) | 1 year
  Target vessel failure (TVF) composite of death, nonfatal myocardial infarction (MI), or ischemic-driven Target Vessel Revascularization (TVR) at 12 months after the procedure.

SECONDARY OUTCOMES:
All death | 1-,6-, and 12-months, and 3-,5-years
Cardiac death | 1-,6-, and 12-months, and 3-,5-years
Myocardial infarction | 1-,6-, and 12-months, and 3-,5-years
Composite of death or myocardial infarction | 1-,6-, and 12-months, and 3-,5-years
Composite of cardiac death or myocardial infarction | 1-,6-, and 12-months, and 3-,5-years
Target-lesion revascularization (TLR) | 1-,6-, and 12-months, and 3-,5-years
Target-vessel revascularization (TVR) | 1-,6-, and 12-months, and 3-,5-years
Stent thrombosis | 1-,6-, and 12-months, and 3-,5-years
  according to Academic Research Consortium (ARC) criteria
Stroke | 1-,6-, and 12-months, and 3-,5-years
Procedural success | 7 days
  Post-procedural diameter stenosis < 30% without death, Q-wave myocardial infarction, or urgent revascularization during the index admission

CONTACTS AND LOCATIONS:
Locations (8):
- South Korea (8):
  - Soon Chun Hyang University Hospital Bucheon, Bucheon-si
  - Daegu Catholic University Medical Center, Daegu
  - Chungnam National University Hospital, Daejeon
  - The Catholic University of Korea, Daejeon ST. Mary's Hospital, Daejeon
  - Chonnam National University Hospital, Gwangju
  - Inje University Pusan Paik Hospital, Pusan
  - Bundang CHA Hospital, Seongnam
  - Asan Medical Center, Seoul

IPD SHARING:
Plan to Share IPD: Undecided